CLINICAL TRIAL: NCT03794401
Title: Alternations of Intestinal Microbiota and Health Impact in Chronic Kidney Disease (AIM-HI CKD): A Cohort Study
Brief Title: Alternations of Intestinal Microbiota and Health Impact in CKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Szu-Chun Hung, Attending physician, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 07-XD-074
Record Dates: First submitted 2019-01-01; First posted 2019-01-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Disease
Keywords: body composition; chronic kidney disease; dietary pattern; gut microbiot
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed to evaluate the impact of dietary pattern, gut microbiota and their interactions on clinical outcomes among patient with CKD stage 3-5.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD stage 3-5 defined as eGFR <60 ml/min/1.73 m2 calculated with the use of the four-variable Modification of Diet in Renal Disease formula who have not yet on dialysis therapy.

Exclusion Criteria:

* Patients with active cancer
* Patients with liver cirrhosis
* Patients have taken antibiotics within three months before screening for inclusion.
* Patients with a cardiac pacemaker or metallic implants,
* Patients are amputees
* Pregnant women
* Patients with inherited renal diseases

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Regional Hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
renal outcome | 3-year follow-up
  a composite of ≥40% decrease in eGFR and ESRD needing chronic dialysis or preemptive kidney transplantation
cardiovascular outcome | 3-year follow-up
  a composite of major adverse CV events, defined as CV death, myocardial infarction, or ischemic stroke

SECONDARY OUTCOMES:
all-cause mortality | 3-year follow-up
  CV death or non-CV death
neurological outcome | 3-year follow-up
  the change of cognitive function or they development of dementia assessed by the Modified Mini-Mental Status Exam annually for 3 years

OTHER OUTCOMES:
change of lean body mass, measured by bioimpedance spectroscopy every 3 months for 2 years | 2-year
  the change of lean body mass

CONTACTS AND LOCATIONS:
Overall Officials: SZU-CHUNG HUNG, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan